CLINICAL TRIAL: NCT05525702
Title: Effects of Multi-model Virtual Reality Intervention Method to Reduce the Prevalence of Delirium in ICU Patients with Mechanical Ventilation
Brief Title: VR Interventions to Reduce the Prevalence of Delirium in ICU Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K4774
Record Dates: First submitted 2022-07-31; First posted 2022-09-01 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Delirium
Keywords: ICU; Virtual Reality; Delirium; family support
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VRFS Intervention (Experimental): Participants will receive standard ICU care and will also undergo VRFS intervention.
  Interventions: Device: VRFS
- Standard ICU Care (No Intervention): Patients will be treated with standard ICU care and not receive VR stimulation.

INTERVENTIONS:
Device: VRFS — Participants wear VR headsets and experience immersive virtual environments, where their family members will be present and offer companionship and comfort.
  Arms: VRFS Intervention

SUMMARY:
The goal of this clinical trial is to learn the effect of VR-based Family Support System (VRFS) on reducing delirium in ICU mechanically ventilated patients. The main question it aims to answer is:

·Using VRFS for participant intervention, can it reduce the incidence of delirium and improve clinical outcomes?

Researchers will investigate whether the implementation of VRFS can reduce the number of delirium days and improve clinical outcomes.

Participants will:

* Receive the VRFS intervention until the endotracheal tube (ETT) is removed.
* Have physiological data collected, including EEG, oxygen saturation levels, ECG, and blood pressure.
* Keep a diary of delirium, dosage of sedative and analgesic drugs, the duration of mechanical ventilation, and ICU stays.

DETAILED DESCRIPTION:
During the VRFS interventions, researchers will fit participants with a VR headset and noise-canceling headphones, shielding them from the ICU environment while allowing family members to be present and offer companionship and comfort.

ELIGIBILITY:
Inclusion Criteria

* Mechanical ventilation duration is expected to be greater than 24 hours;
* ICU stay duration is expected to be greater than 72 hours;
* Age is 18 years or older, with no upper age limit;
* Language: Chinese. Exclusion Criteria
* Severe visual or auditory impairments (diplopia, low vision due to macular degeneration, retinopathy; severe hearing loss or deafness);
* Cognitive and consciousness disturbances prior to ICU admission;
* Severe motion sickness;
* Head trauma or surgery that prevents the wearing of equipment;
* A history of long-term use of antipsychotic and/or benzodiazepine medications.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Delirium Day | 2 years
  Delirium is monitored and evaluated by the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). The CAM-ICU has four items ((1) altered mental status/fluctuating course, (2)inattention, (3) altered level of consciousness, and (4) disorganized thinking) and each item has two factors (positive or negative). The physicians can diagnose the patients with delirium when the results of item (1), item (2), and item (3) or item (4) are positive.

SECONDARY OUTCOMES:
ICU Days | 2 years
  The ICU stays are daily recorded by the physicians and nurses in ICU.
Duration of Mechanical Ventilation | 2 years
  The duration of mechanical ventilation is daily recorded by the physicians and nurses.
Electroencephalogram (EEG) | 2 years
  A wearable headset device was utilized to obtain consistent and adequate quality EEG data.
Oxygen saturation level | 2 years
  The oxygen saturation level (SpO2, %) will be collected from a bedside monitor before the intervention.
Blood pressure | 2 years
  The blood pressure(mmHg) will be collected from a bedside monitor after the intervention. Both Systolic and Diastolic Blood Pressure will be measured.
Dosage of sedative and analgesic drugs | 2 years
  Daily records by doctors and nurses.

CONTACTS AND LOCATIONS:
Overall Officials: Yun Long, MD, Study Director — Peking Union Medical College
Locations (1):
- PUMC, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nassar Junior AP, Besen BAMP, Robinson CC, Falavigna M, Teixeira C, Rosa RG. Flexible Versus Restrictive Visiting Policies in ICUs: A Systematic Review and Meta-Analysis. Crit Care Med. 2018 Jul;46(7):1175-1180. doi: 10.1097/CCM.0000000000003155. PMID 29642108
- [Background] da Silva Ramos FJ, Fumis RR, Azevedo LC, Schettino G. Perceptions of an open visitation policy by intensive care unit workers. Ann Intensive Care. 2013 Oct 17;3(1):34. doi: 10.1186/2110-5820-3-34. PMID 24135292
- [Background] Mohsen S, Moss SJ, Lucini F, Krewulak KD, Stelfox HT, Niven DJ, Sauro KM, Fiest KM. Impact of Family Presence on Delirium in Critically Ill Patients: A Retrospective Cohort Study. Crit Care Med. 2022 Nov 1;50(11):1628-1637. doi: 10.1097/CCM.0000000000005657. Epub 2022 Aug 26. PMID 36044306
- [Background] Deng LX, Cao L, Zhang LN, Peng XB, Zhang L. Non-pharmacological interventions to reduce the incidence and duration of delirium in critically ill patients: A systematic review and network meta-analysis. J Crit Care. 2020 Dec;60:241-248. doi: 10.1016/j.jcrc.2020.08.019. Epub 2020 Aug 31. PMID 32919363
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Background] van den Boogaard M, Schoonhoven L, Evers AW, van der Hoeven JG, van Achterberg T, Pickkers P. Delirium in critically ill patients: impact on long-term health-related quality of life and cognitive functioning. Crit Care Med. 2012 Jan;40(1):112-8. doi: 10.1097/CCM.0b013e31822e9fc9. PMID 21926597
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Mehta S, Cook D, Devlin JW, Skrobik Y, Meade M, Fergusson D, Herridge M, Steinberg M, Granton J, Ferguson N, Tanios M, Dodek P, Fowler R, Burns K, Jacka M, Olafson K, Mallick R, Reynolds S, Keenan S, Burry L; SLEAP Investigators; Canadian Critical Care Trials Group. Prevalence, risk factors, and outcomes of delirium in mechanically ventilated adults. Crit Care Med. 2015 Mar;43(3):557-66. doi: 10.1097/CCM.0000000000000727. PMID 25493968
- [Background] Wiegand TLT, Remi J, Dimitriadis K. Electroencephalography in delirium assessment: a scoping review. BMC Neurol. 2022 Mar 11;22(1):86. doi: 10.1186/s12883-022-02557-w. PMID 35277128
- [Background] Salluh JI, Soares M, Teles JM, Ceraso D, Raimondi N, Nava VS, Blasquez P, Ugarte S, Ibanez-Guzman C, Centeno JV, Laca M, Grecco G, Jimenez E, Arias-Rivera S, Duenas C, Rocha MG; Delirium Epidemiology in Critical Care Study Group. Delirium epidemiology in critical care (DECCA): an international study. Crit Care. 2010;14(6):R210. doi: 10.1186/cc9333. Epub 2010 Nov 23. PMID 21092264
- [Background] Janssen TL, Alberts AR, Hooft L, Mattace-Raso F, Mosk CA, van der Laan L. Prevention of postoperative delirium in elderly patients planned for elective surgery: systematic review and meta-analysis. Clin Interv Aging. 2019 Jun 19;14:1095-1117. doi: 10.2147/CIA.S201323. eCollection 2019. PMID 31354253
- [Background] Chen H, Mo L, Hu H, Ou Y, Luo J. Risk factors of postoperative delirium after cardiac surgery: a meta-analysis. J Cardiothorac Surg. 2021 Apr 26;16(1):113. doi: 10.1186/s13019-021-01496-w. PMID 33902644
- [Background] Thom RP, Levy-Carrick NC, Bui M, Silbersweig D. Delirium. Am J Psychiatry. 2019 Oct 1;176(10):785-793. doi: 10.1176/appi.ajp.2018.18070893. No abstract available. PMID 31569986